CLINICAL TRIAL: NCT00591760
Title: Correction of Growth Hormone Deficiency in Patients With Chronic Heart Failure: a Randomized, Controlled, Single-blind Study
Brief Title: Growth Hormone Deficiency in Chronic Heart Failure: A Preliminary Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Antonio Cittadini, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GH replacement in CHF
Record Dates: First submitted 2007-12-20; First posted 2008-01-11 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2009-03

CONDITIONS: Heart Failure; Growth Hormone Deficiency; Ischemic Heart Disease
Keywords: Heart Failure; Growth Hormone; Anabolism; Anabolic Deficiency; Hormone replacement
MeSH Terms: conditions — Heart Failure; Dwarfism, Pituitary; Myocardial Ischemia | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GH (Experimental): Patients will receive 6 months of substitutive somatotropin (growth hormone) therapy at a dose of 0.012 mg/kg every second day, added to their background optimized CHF therapy
  Interventions: Drug: Somatotropin
- Placebo (No Intervention): PLacebo will be admistred with the same devices of GH, also on top of Optimal CHF treatment

INTERVENTIONS:
Drug: Somatotropin — Subcutaneous Somatotropin (recombinant human Growth Hormone) 0.012 mg/kg every second day for 6 months
  Other Names: rhGH; Saizen; NutropinAq
  Arms: GH

SUMMARY:
The aim of this study is to investigate the potential benefits of the correction of growth hormone (GH) deficiency with GH replacement therapy in patients with chronic heart failure due to left ventricular systolic dysfunction.

DETAILED DESCRIPTION:
To date, a wide range of alterations in the GH/IGF-1 axis have been described in patients with chronic heart failure (CHF): reductions in GH levels, reductions in IGF-1 and a pattern of peripheral resistance to GH, in particular in patients with severe heart failure and cardiac cachexia. Unpublished experience of our group support the concept that a considerable amount of CHF-patients have a coexisting Growth Hormone Deficiency (GHD), defined by current guidelines(GH stimulation test).

Our study hypothesis is that correction of GH deficiency in patients with chronic heart failure may exert a beneficial effect on their cardiac function and remodeling, performance status and quality-of-life.

Since this was a preliminary study, no sample size calculation was performed; treatment effects from were sought in left ventricular function (as assessed by cardiac MRI), cardiopulmonary exercise performance, clinical status, vascular reactivity, biochemistry and neurohumoral markers of disease (NT-proBNP).

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure in ew York Heart Association functional class II to IV
* Left ventricular end diastolic diameter > 60 mm
* Left ventricular ejection fraction < 40%
* Growth Hormone Deficiency (defined as a peak GH response to intravenous stimulation with GHRH + Arginine < 9 ng/dl)
* Age 18-80 years
* Clinical stability, guideline-oriented maximal pharmacological therapy
* Informed consent

Exclusion Criteria:

* Active Myocarditis
* Hypertrophic Cardiomyopathy
* Active endocarditis
* Active malignancy
* End stage renal disease
* Severe liver disease (Child B-C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cittadini, MD, Principal Investigator — Federico II University - Naples; Luigi Saccà, MD, Study Chair — Federico II University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-three patients with CHF NYHA class II-IV and GH deficiency were enrolled from December 2004 to December 2006. These patients were consecutively selected from a cohort of 158 ambulatory patients referred to our tertiary care center and, to a minor extent, patients hospitalized for CHF.
Pre-assignment Details: Patients recruited during hospital stay were studied after a 3-months period of optimized medical therapy and clinical stability
Groups:
- GH Replacement Therapy: Patients will receive 6 months of substitutive somatotropin (growth hormone) therapy at a dose of 0,00415 mg/kg a day, added to their background optimized CHF therapy
- Control: Optimal CHF treatment
Period: Overall Study
Arm/Group | GH Replacement Therapy | Control
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GH Replacement Therapy | Control | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 15 | 17 | 32.0
  >=65 years | 13 | 11 | 24.0
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (6) | 62 (8) | 62 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9.0
  Male | 24 | 23 | 47.0
echocardiography [Mean (Full Range); unit: % of ejection fraction] | 30 [20 to 70] | 40 [20 to 70] | 35 [20 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2
Description: changes in peak VO2
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ml/kg/min
Arm/Group | GH Replacement Therapy | Control
Number analyzed (Participants) | 28 | 28
ml/kg/min | 14.5 (1.0) | 12.9 (1.0)

ADVERSE EVENTS:
Arm/Group | GH Replacement Therapy | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No